CLINICAL TRIAL: NCT03628755
Title: Effectiveness of Digital Manipulation of Thyroid Cartilage and Fluency Shaping Therapy for the Management of Stuttering in Adult
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Isra University (Other)
Responsible Party: Principal Investigator, Nasir Khan, Research Associate, Isra University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IIRS-IUISB/PHD/016
Record Dates: First submitted 2018-08-09; First posted 2018-08-14 (Actual); Last update posted 2019-07-26 (Actual); Status verified 2019-07

CONDITIONS: Developmental Stuttering
Keywords: Fluency shaping therapy; Digital Manipulation; Stuttering; communication
MeSH Terms: conditions — Stuttering; Communication

STUDY DESIGN:
Intervention Model Description: The three group were digital manipulation of thyroid cartilage(DMT) group,fluency shaping therapy (FST) group,combination of DMT,FST. the intervention period for each subject was three month and data was collected on day one and at the end of every 2 weeks. 4th week , 8th week, and 12th week which were aimed to reduce severity of stuttering and improve fluency
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Digital Manipulation (Active Comparator): Digital manipulation of thyroid cartilage (DMT) Duration: Each child was given 15-20 minute session. Frequency: Twice in a week. Total 24 sessions were performed. The aim of DMT was to reduce the severity of stuttering and improve the fluency.
  Interventions: Behavioral: Digital Manipulation of Thyroid cartilage
- fluency shaping Therapy (Active Comparator): Fluency Shaping Therapy Duration:Each child was given 30-minute session. Fluency Shaping Therapy (FST) Frequency: Twice in a week Total 24 sessions were performed.
  The aim of DMT was to reduce the severity of stuttering and improve the fluency
  Interventions: Behavioral: Fluency Shaping Therapy
- combination Group (Experimental): Combination Group (DMT+FST) Duration:Each subject was given 45-Minute session Frequency: Twice in a week Total 24 sessions were performed combination group was more significant option for reducing the severity of stuttering and improve fluency than practice the single DMT or FST
  Interventions: Behavioral: Digital Manipulation of Thyroid cartilage; Behavioral: Fluency Shaping Therapy; Behavioral: combination Group

INTERVENTIONS:
Behavioral: Digital Manipulation of Thyroid cartilage — Digital manipulation of thyroid cartilage was applied to the anterior aspect of thyroid cartilage while using the thumb or finger and the patient was asked to speak.
  prolongation of vowel is 7 to 8 seconds, voice rest after each set is 10 second.
  total repetition is 60.
  Arms: Digital Manipulation; combination Group
Behavioral: Fluency Shaping Therapy — FST session comprised of speech techniques such as prolongation of sounds, easy onset, continuous phonation, light articulatory contact, in reading and conversation in three speaking situations (speaking with therapist, reading aloud, and free conversation Reading task was for 80 short phrases.
  Arms: combination Group; fluency shaping Therapy
Behavioral: combination Group — combination group intervention of DMT + FST
  Arms: combination Group

SUMMARY:
This study was conducted to determine the effectiveness of digital manipulation of thyroid cartilage for the management of stuttering in adult.There were three groups,Group A received Digital Manipulation of Thyroid cartilage (DMT),Group B received Fluency shaping Therapy(FST),Group C received combination of DMT,FST.

DETAILED DESCRIPTION:
The purpose of speech therapy is to stop progression of stuttering while teaching the method to client how to cope efficiently his or her stuttering disorder.

The goal of fluency shaping therapy to eliminate the severity of stuttering by adopting the specific pattern of speech production and also reduce negative reaction to stuttering by default).

Digital manipulation of thyroid cartilage decreases tension in vocal fold and reduces severity of stuttering and improves production of speech. DMT reduces unnecessary amount of tension in vocal tract and participant speaks with relax respiration,phonation, articulation and facilitate more fluent.in DMT subject speaks in natural way rather than in specific method in every situation.

ELIGIBILITY:
Inclusion Criteria:

* Developmental stuttering
* Between age of 18 to 30 years
* Only male

Exclusion Criteria:

* Language disorders
* Cluttering
* Neurological stuttering

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-07-18 (Actual)

PRIMARY OUTCOMES:
Scale for Rating the severity of stuttering | 12 weeks
  0-No Stuttering
  1. Very mild-stuttering .
  2. Mild-stuttering.
  3. Mild to moderate-stuttering.
  4. Moderate -stuttering.
  5. Moderate to severe stuttering
  6. Severe-stuttering . 7 Very severe -stuttering .
Modified Erickson scale of communication attitude(24) | 12week
  This 24-item scale distinguishes the extent to which a stuttering person's communication attitude deviates from normed attitudes. Statement require a true or false answer. Individual with mean score of 19.22 and range of 9-24 is consider as stutter. Individual with mean score of 9.4 and range of 1-21 is consider as non-stutter. The higher the score, the poorer the communication attitude.
Assessment of Physiological Factors Associated with Stuttering | 12 week
  Clinician need to carefully observe whether these physiological factor are present or not present during stuttering. 0=not present 1= present

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Rehabilitation Medicine (NIRM), Islamabad, Federal, Pakistan